CLINICAL TRIAL: NCT01467843
Title: Comparison of CAM and Conventional Mind-Body Therapies for Chronic Back Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R01AT006226-01A1 (NIH)
Record Dates: First submitted 2011-11-07; First posted 2011-11-09 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Low Back Pain
Keywords: Cognitive Behavioral Therapy; Mindfulness Based Stress Reduction
MeSH Terms: conditions — Low Back Pain | interventions — Cognitive Behavioral Therapy; Mindfulness-Based Stress Reduction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cognitive Behavioral Therapy (Active Comparator): Participants randomized to the CBT intervention will attend eight weekly 2 hour sessions.
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Mindfulness-Based Stress Reduction (Active Comparator): Participants randomized to the MBSR arm will attend eight weekly 2 hour MBSR sessions.
  Interventions: Behavioral: Mindfulness Based Stress Reduction
- Usual Care (No Intervention): Participants randomized to Usual Care will continue to receive care for their low back pain as prescribed by his/her Primary Care Physician.

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — The Cognitive Behavioral Therapy Intervention will be delivered during 8 weekly classes each lasting 2 hours. The classes will be held at a conveniently located Group Health Facility.
  Arms: Cognitive Behavioral Therapy
Behavioral: Mindfulness Based Stress Reduction — The Mindfulness Based Stress Reduction Classes will be delivered in 8 weekly classes each lasting 2 hours.
  Arms: Mindfulness-Based Stress Reduction

SUMMARY:
Although national expenditures on back pain treatments have increased substantially over the past decade, the health and functional status of persons suffering from back pain has deteriorated. This trial will evaluate the effectiveness, and cost-effectiveness, of a safe and relatively inexpensive "mind-body" therapy that has the potential to provide relief to some of the millions of Americans who continue to suffer from chronic back pain.

DETAILED DESCRIPTION:
Chronic back pain remains one of the most common and challenging public health problems in the U.S.. Although the amount of money spent on back pain treatments has increased substantially over the past decade in the U.S., the health and functional status of persons suffering from back pain has deteriorated. There is a clear need to identify safe, effective, and cost-effective treatment options for this often debilitating and expensive problem. Some of the more promising treatments for chronic back pain include "mind-body" therapies that address both psychological and somatic aspects of the pain experience. This randomized trial will compare the effectiveness and cost-effectiveness of Mindfulness-Based Stress Reduction (MBSR), a well-established but inadequately-studied CAM mind-body therapy, with usual care for persons with chronic low back pain and dysfunction. This trial will also compare MBSR with a conventional mind-body therapy, Cognitive-Behavioral Therapy (CBT), which has been found to be a modestly to moderately effective treatment for chronic back pain. Should MBSR and/or CBT prove effective in this trial, the mechanisms (mediators) of the effects of these two different mind-body therapies on pain and dysfunction will be explored. Because CBT aims to alter patients' cognitive and behavioral responses to pain, whereas MBSR focuses on direct present moment experience and not on changing the thoughts or feelings about such experience, these two therapies are hypothesized to operate by different mechanisms. A total of 342 adults aged 20 through 70 years who have moderately to severely disabling chronic back pain will be recruited and randomized in equal proportions to MBSR, CBT, and treatment as usual (usual care). Both the MBSR and CBT interventions will be provided to groups of up to 15 participants once a week for 8 weeks. The primary outcomes will be back pain-related functional limitations (Roland scale) and pain bothersomeness (rated on a 0-10 scale). Secondary outcomes include depression, anxiety, perceived stress, pain interference with activities, and sleep disturbance. Outcomes will be measured 4, 8, 26, and 52 weeks after randomization. If MBSR is at least moderately more effective than usual care, this safe and relatively inexpensive therapy would provide an appealing treatment option for chronic back pain that could be made more widely available. Because of the high prevalence and costs of chronic back pain, treatments with even modest impact on pain and function could produce a large benefit on a population level.

ELIGIBILITY:
Inclusion Criteria:

* clinical Diagnosis of Low Back Pain lasting at least 3 months
* pain of at least 4 on a 0-10 bothersomeness scale

Exclusion Criteria:

* do not currently have back pain
* current back pain episode less then 3 months in duration
* current back pain is only reported as mild in dysfunction and symptoms (i.e., less than a score of 7 on the 0-23 modified Roland Scale or a bothersomeness score lower than 4 on a 0-10 scale);
* sciatica
* underlying systemic or visceral disease
* pregnancy
* abdominal aneurisms
* spondylolisthesis
* discitis
* spinal stenosis
* spinal infections
* cancer or unexplained weight loss
* recent vertebral fracture
* current or past participation in classes or therapies closely resembling our MBSR or CBT interventions for chronic pain
* have physical problems that won't allow them to do yoga (i.e., gross obesity, severe pain when bending or twisting, unable to get up and down from the floor)
* involved with litigation or compensation claim for back pain
* evidence of severe or progressive neurologic deficits
* radiculopathy
* fibromyalgia diagnosis
* rheumatoid arthritis
* back surgery within the last 2 years
* unstable medical or severe psychiatric conditions
* unable to speak or read English
* unable to hear
* plan to move out of town

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 342 (Actual)
Dates: Start 2012-06; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Back pain-related dysfunction | 26 weeks
  Back-related dysfunction will be measured with the modified Roland Disability Questionnaire ("Roland scale"), which asks whether 23 specific activities were limited due to back pain during the past week (yes or no). This measure has been found to be reliable, valid and sensitive to clinical changes and is appropriate for telephone administration and patients with moderate disability.
Bothersomeness of back pain | 26 weeks
  Symptom bothersomeness will be measured by asking participants to rate how "bothersome" their back pain has been during the previous week on a 0 to 10 scale (0 = "not at all bothersome" and 10 = "extremely bothersome"). This question worked well in our previous trials and is highly correlated with a 0-10 measure of pain intensity (r=0.8 to 0.9). It is also highly correlated with measures of function and other outcome measures.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Cherkin, PhD, Principal Investigator — Kaiser Permanente
Locations (1):
- Group Health Cooperative, Seattle, Washington, United States

REFERENCES:
- [Derived] Chen JA, Anderson ML, Cherkin DC, Balderson BH, Cook AJ, Sherman KJ, Turner JA. Moderators and Nonspecific Predictors of Treatment Benefits in a Randomized Trial of Mindfulness-Based Stress Reduction vs Cognitive-Behavioral Therapy vs Usual Care for Chronic Low Back Pain. J Pain. 2023 Feb;24(2):282-303. doi: 10.1016/j.jpain.2022.09.014. Epub 2022 Sep 28. PMID 36180008
- [Derived] Cherkin DC, Sherman KJ, Balderson BH, Cook AJ, Anderson ML, Hawkes RJ, Hansen KE, Turner JA. Effect of Mindfulness-Based Stress Reduction vs Cognitive Behavioral Therapy or Usual Care on Back Pain and Functional Limitations in Adults With Chronic Low Back Pain: A Randomized Clinical Trial. JAMA. 2016 Mar 22-29;315(12):1240-9. doi: 10.1001/jama.2016.2323. PMID 27002445
- [Derived] Cherkin DC, Sherman KJ, Balderson BH, Turner JA, Cook AJ, Stoelb B, Herman PM, Deyo RA, Hawkes RJ. Comparison of complementary and alternative medicine with conventional mind-body therapies for chronic back pain: protocol for the Mind-body Approaches to Pain (MAP) randomized controlled trial. Trials. 2014 Jun 7;15:211. doi: 10.1186/1745-6215-15-211. PMID 24906419